CLINICAL TRIAL: NCT03491553
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Safety, Tolerability and Antiviral Activity of GS-9688 in Virally-Suppressed Adult Subjects With Chronic Hepatitis B
Brief Title: Safety, Tolerability and Antiviral Activity of Selgantolimod in Virally-Suppressed Participants With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-389-2024; ACTRN12618000143224p (Registry Identifier: ANZCTR)
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — selgantolimod; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Selgantolimod 3 mg: HBeAg-positive CHB Participants (Experimental): Participants with Hepatitis B e Antigen (HBeAg)-positive CHB will remain on their current OAV and receive selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/early discontinuation (ED). At Week 48, per Principal Investigator's (PI's) discretion, participants can continue in the Treatment Free Follow-Up (TFFU) phase for up to an additional 48 weeks.
  Interventions: Drug: Selgantolimod; Drug: Hepatitis B virus (HBV) OAV Therapy
- Selgantolimod 3 mg: HBeAg-negative CHB Participants (Experimental): Participants with HBeAg-negative CHB will remain on their current OAV and receive selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Selgantolimod; Drug: Hepatitis B virus (HBV) OAV Therapy
- Selgantolimod 1.5 mg: HBeAg-positive CHB Participants (Experimental): Participants with HBeAg-positive CHB will remain on their current OAV and receive selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Selgantolimod; Drug: Placebo; Drug: Hepatitis B virus (HBV) OAV Therapy
- Selgantolimod 1.5 mg: HBeAg-negative CHB Participants (Experimental): Participants with HBeAg-negative CHB will remain on their current OAV and receive selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Selgantolimod; Drug: Placebo; Drug: Hepatitis B virus (HBV) OAV Therapy
- Placebo: HBeAg-positive CHB Participants (Experimental): Participants with HBeAg-positive CHB will remain on their current OAV and receive 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Placebo; Drug: Hepatitis B virus (HBV) OAV Therapy
- Placebo: HBeAg-negative CHB Participants (Experimental): Participants with HBeAg-negative CHB will remain on their current OAV and receive 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants will continue their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants can continue in the TFFU phase for up to an additional 48 weeks.
  Interventions: Drug: Placebo; Drug: Hepatitis B virus (HBV) OAV Therapy

INTERVENTIONS:
Drug: Selgantolimod — Tablet(s) administered orally once weekly
  Other Names: GS-9688
  Arms: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants; Selgantolimod 1.5 mg: HBeAg-positive CHB Participants; Selgantolimod 3 mg: HBeAg-negative CHB Participants; Selgantolimod 3 mg: HBeAg-positive CHB Participants
Drug: Placebo — Placebo to match (PTM) selgantolimod tablet(s) administered orally once weekly
  Arms: Placebo: HBeAg-negative CHB Participants; Placebo: HBeAg-positive CHB Participants; Selgantolimod 1.5 mg: HBeAg-negative CHB Participants; Selgantolimod 1.5 mg: HBeAg-positive CHB Participants
Drug: Hepatitis B virus (HBV) OAV Therapy — Commercially available HBV OAV therapy could include one of the following:
  Tenofovir disoproxil fumarate (TDF; Viread®) Entecavir (Baraclude®) Adefovir (Hepsera®) Lamivudine (Epivir® ) Telbivudine (Tyzeka®) Tenofovir alafenamide (TAF; Vemlidy®)

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability and antiviral activity of selgantolimod (formerly GS-9688) in virally suppressed chronic hepatitis B (CHB) adults on oral antiviral (OAV) agents.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Adult males and non-pregnant, non-lactating females
* Documented evidence of chronic HBV infection with detectable hepatitis B surface antigen (HBsAg) levels
* On commercially available HBV OAV treatment(s) for at least 6 months with no change in regimen for 3 months prior to screening
* HBV Deoxyribonucleic acid (DNA) ≤ 20 IU/mL for 6 or more months prior to screening
* Screening Electrocardiogram (ECG) without clinically significant abnormalities

Key Exclusion Criteria:

* Extensive bridging fibrosis or cirrhosis
* Adults meeting any of the protocol defined exclusionary laboratory parameters at screening:

  * Alanine aminotransferase (ALT) > 3x Upper Limit of Normal (ULN)
  * International normalized ratio (INR) > ULN unless the adult is stable on an anticoagulant regimen
  * Albumin < 3.5 g/dL
  * Direct bilirubin > 1.5x ULN
  * Platelet Count < 100,000/uL
  * Estimated creatinine clearance < 60 mL/min (using the Cockcroft-Gault method)
* Co-infection with human immunodeficiency virus, hepatitis C virus or hepatitis D virus
* Prior history of hepatocellular carcinoma (HCC) or screening alpha-fetoprotein ≥ 50 ng/mL without imaging
* Diagnosis of autoimmune disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease, hemoglobinopathy, retinal disease, or are immunosuppressed.
* Chronic liver disease of a non-HBV etiology, except for non-alcoholic fatty liver disease
* Received solid organ or bone marrow transplant
* Received prolonged therapy with immunomodulators or biologics within 3 months of screening
* Use of another investigational agent within 90 days of screening, unless allowed by the Sponsor

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States
- Auckland Clinical Studies Limited, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brooks AE, Verdon D, Eom J, Ng J, Steemson H, Lau AH, et al. Peripheral Immune Responses to Toll-Like Receptor 8 Agonist Selgantolimod (GS-9688) in Patients with Chronic Hepatitis B [Poster]. AASLD: The Liver Meeting® 2019; 2019 08-12 November; Boston, MA.
- [Result] Gane E, Zhao Y, Tan SK, Lau AH, Gaggar A, Subramanian M, et al. Efficacy and Safety of Oral TLR8 Agonist Selgantolimod in Virally Suppressed Adult Patients With Chronic Hepatitis B: a Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study [Poster 697]. AASLD: The Liver Meeting® 2019; 2019 08-12 November; Boston, MA.
- [Result] Chen DY, C. M, Tan SK, Yang JC, Gane EJ, Janssen HLA, et al. Characterization of Cytokine Response to Toll-Like Receptor 8 Agonist Selgantolimod in Viremic and Virally Suppressed Chronic Hepatitis B Patients [Poster 0721]. American Association for the Study of Liver Diseases (AASLD): The Liver Meeting Digital Experience; 2020 13-16 November.
- [Result] Chen D, Kim S, Brooks A, McDonald C, Yang J, Gaggar A, et al. Potential Biomarkers of Response in Chronic Hepatitis B Patients Who Achieved HBeAg Loss Upon Treatment With Toll-Like Receptor 8 Agonist Selgantolimod [Poster FR1350]. The Digital International Liver Congress (ILC); 2020 27-29 August.
- [Result] Gane E, Dubar PR, Brooks AE, Zhao Y, Tan SK, Lau AH, et al. Efficacy and Safety of 24 Weeks Treatment with Oral TLR8 Agonist Selgantolimod (GS-9688, SLGN) in Virally Suppressed Adult Patients with Chronic Hepatitis B: A Phase 2 Study [Presentation]. The Digital International Liver Congress (ILC); 2020 27-29 August.
- [Derived] Gane EJ, Dunbar PR, Brooks AE, Zhang F, Chen D, Wallin JJ, van Buuren N, Arora P, Fletcher SP, Tan SK, Yang JC, Gaggar A, Kottilil S, Tang L. Safety and efficacy of the oral TLR8 agonist selgantolimod in individuals with chronic hepatitis B under viral suppression. J Hepatol. 2023 Mar;78(3):513-523. doi: 10.1016/j.jhep.2022.09.027. Epub 2022 Oct 29. PMID 38133554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in New Zealand and the United States. The first participant was screened on 6 April 2018. The last study visit occurred on 10 August 2020.
Pre-assignment Details: 59 participants were screened.
Groups:
- Selgantolimod 3 mg: HBeAg-positive CHB Participants: Participants with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B (CHB) remained on their current oral antiviral (OAV) and received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/early discontinuation (ED). At Week 48, per Principal Investigator's (PI's) discretion, participants could continue in the Treatment Free Follow-Up (TFFU) phase for up to an additional 48 weeks.
- Selgantolimod 3 mg: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
- Selgantolimod 1.5 mg: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
- Selgantolimod 1.5 mg: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
- Placebo: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
- Placebo: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
Period: Main Study (Up to Week 48)
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Started | 9 | 10 | 10 | 10 | 5 | 4
Completed | 8 | 9 | 10 | 9 | 5 | 4
Not Completed | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew Consent | 1 | 1 | 0 | 0 | 0 | 0
Period: TFFU (Week 49 up to Additional 48 Weeks)
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Started | 0 (8 participants completed the study period up to Week 48 but did not continue in the TFFU phase.) | 1 (9 participants completed the study period up to Week 48 but only 1 participant continued in the TFFU phase.) | 0 (10 participants completed the study period up to Week 48 but did not continue in the TFFU phase.) | 0 (9 participants completed the study period up to Week 48 but did not continue in the TFFU phase.) | 0 (5 participants completed the study period up to Week 48 but did not continue in the TFFU phase.) | 0 (4 participants completed the study period up to Week 48 but did not continue in the TFFU phase.)
Completed | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who took at least 1 dose of the study drug.
Groups:
- Selgantolimod 3 mg: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED. At Week 48, per PI's discretion, participants could continue in the TFFU phase for up to an additional 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants | Total
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7.8) | 46 (10.1) | 43 (5.6) | 53 (6.8) | 43 (7.9) | 57 (10.5) | 47 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 1 | 2 | 12
  Male | 7 | 7 | 7 | 9 | 4 | 2 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 10 | 10 | 5 | 4 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 6 | 5 | 7 | 3 | 2 | 28
  Black or African American | 0 | 3 | 0 | 1 | 0 | 1 | 5
  Native Hawaiian or Pacific Islander | 4 | 1 | 4 | 1 | 1 | 1 | 12
  White | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 7 | 1 | 6 | 0 | 2 | 17
  New Zealand | 8 | 3 | 9 | 4 | 5 | 2 | 31
Hepatitis B Surface Antigen (HBsAg) [Mean (Standard Deviation); unit: log10 IU/mL] | 3.4 (0.57) | 2.6 (1.58) | 3.4 (0.62) | 1.7 (1.10) | 3.3 (0.46) | 3.2 (0.42) | 2.9 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum Quantitative Hepatitis B Surface Antigen (qHBsAg) From Baseline at Week 24
Time Frame: Week 24
Population: The Full Analysis Set included all randomized participants who took at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Selgantolimod 3 mg: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
- Selgantolimod 3 mg: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received selgantolimod 3 mg (2 x 1.5 mg tablet) orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
- Selgantolimod 1.5 mg: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
- Selgantolimod 1.5 mg: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received selgantolimod 1.5 mg (1 x 1.5 mg tablet) plus 1 tablet of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
- Placebo: HBeAg-positive CHB Participants: Participants with HBeAg-positive CHB remained on their current OAV and received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
- Placebo: HBeAg-negative CHB Participants: Participants with HBeAg-negative CHB remained on their current OAV and received 2 tablets of placebo orally on the same day once a week (every 7 days) for 24 doses. After the 24th dose, participants continued their current OAV therapy until Week 48/ED.
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 10.0 [0.3 to 44.5] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
Statistical Analysis 1: Comparison: Selgantolimod 3 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 2: Comparison: Selgantolimod 3 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 3: Comparison: Selgantolimod 1.5 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 4: Comparison: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 10.0, 95% CI 2-sided [-47.2 to 47.1] — The 2-sided 95% CI for the percentage difference by HBeAg status was constructed based on the standardized statistic and inverting two 1-sided tests

2. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
Statistical Analysis 1: Comparison: Selgantolimod 3 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 2: Comparison: Selgantolimod 3 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 3: Comparison: Selgantolimod 1.5 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 4: Comparison: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0

3. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
Statistical Analysis 1: Comparison: Selgantolimod 3 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 2: Comparison: Selgantolimod 3 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 3: Comparison: Selgantolimod 1.5 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 4: Comparison: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0

4. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
Statistical Analysis 1: Comparison: Selgantolimod 3 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 2: Comparison: Selgantolimod 3 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 3: Comparison: Selgantolimod 1.5 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 4: Comparison: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0

5. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in Serum qHBsAg From Baseline at Week 48
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 [0.0 to 33.6] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 10.0 [0.3 to 44.5] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
Statistical Analysis 1: Comparison: Selgantolimod 3 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 2: Comparison: Selgantolimod 3 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 3: Comparison: Selgantolimod 1.5 mg: HBeAg-positive CHB Participants vs Placebo: HBeAg-positive CHB Participants; Test type: Other; Percentage Difference = 0.0
Statistical Analysis 4: Comparison: Selgantolimod 1.5 mg: HBeAg-negative CHB Participants vs Placebo: HBeAg-negative CHB Participants; Test type: Other; Percentage Difference = 10.0, 95% CI 2-sided [-47.2 to 47.1] — [estimate comment as in outcome 1, analysis 4]

6. Secondary Outcome: Change From Baseline in Serum qHBsAg at Week 4
Time Frame: Baseline, Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 7 | 10 | 9 | 10 | 5 | 4
log10 IU/mL | 0.02 (0.047) | -0.07 (0.110) | 0.00 (0.070) | -0.01 (0.127) | -0.02 (0.034) | -0.03 (0.058)

7. Secondary Outcome: Change From Baseline in Serum qHBsAg (log10 IU/mL) at Week 8
Time Frame: Baseline, Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 8 | 10 | 10 | 9 | 5 | 4
log10 IU/mL | 0.00 (0.051) | -0.05 (0.117) | -0.01 (0.041) | -0.04 (0.119) | 0.02 (0.041) | -0.03 (0.061)

8. Secondary Outcome: Change From Baseline in Serum qHBsAg (log10 IU/mL) at Week 12
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 8 | 10 | 10 | 9 | 5 | 4
log10 IU/mL | -0.01 (0.059) | -0.05 (0.117) | 0.00 (0.050) | -0.04 (0.115) | 0.05 (0.034) | 0.00 (0.048)

9. Secondary Outcome: Change From Baseline in Serum qHBsAg (log10 IU/mL) at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 8 | 7 | 8 | 9 | 5 | 4
log10 IU/mL | 0.01 (0.059) | -0.05 (0.136) | -0.05 (0.059) | -0.16 (0.460) | -0.02 (0.048) | -0.01 (0.066)

10. Secondary Outcome: Change From Baseline in Serum qHBsAg (log10 IU/mL) at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 5 | 4
log10 IU/mL | -0.01 (0.073) | -0.05 (0.145) | -0.07 (0.110) | -0.17 (0.523) | 0.00 (0.049) | -0.05 (0.050)

11. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at Week 12
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 | 10.0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 24
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 | 10.0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 48
Description: HBsAg loss was defined as qualitative HBsAg changing from positive at baseline to negative at a postbaseline visit.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 5 | 4
percentage of participants | 0 | 10.0 | 0 | 10.0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 12
Description: HBeAg loss was defined as qualitative HBeAg changing from positive at baseline to negative at a postbaseline visit. HBeAg seroconversion was defined as HBeAb test changing from negative or missing at baseline to positive at a postbaseline visit.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed. Analysis was performed only on HBeAg-positive CHB participants.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Placebo: HBeAg-positive CHB Participants
Number analyzed (Participants) | 9 | 10 | 5
percentage of participants
  HBeAg Loss | 0 | 10.0 | 0
  HBeAg Loss and Seroconversion | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 24
Description: as for outcome 14
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed. Analysis was performed only on HBeAg-positive CHB participants.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Placebo: HBeAg-positive CHB Participants
Number analyzed (Participants) | 9 | 10 | 5
percentage of participants
  HBeAg Loss | 0 | 10.0 | 0
  HBeAg Loss and Seroconversion | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 48
Description: HBeAg loss was defined as qualitative HBeAg changing from positive at baseline to negative at a postbaseline visit. HBeAg seroconversion was defined as hepatitis B e antibody (HBeAb) test changing from negative or missing at baseline to positive at a postbaseline visit.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. Analysis was performed only on HBeAg-positive CHB participants.
Measure: Number; unit: percentage of participants
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Placebo: HBeAg-positive CHB Participants
Number analyzed (Participants) | 9 | 10 | 5
percentage of participants
  HBeAg Loss | 22.2 | 10.0 | 0
  HBeAg Loss and Seroconversion | 11.1 | 0 | 0

17. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Virologic breakthrough was defined as having two consecutive visits of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) ≥ 69 IU/mL.
Time Frame: Baseline up to Week 48
Population: There were no participants analyzed for the outcome measure since none of the participants met the criteria.
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Drug Resistance Mutations
Description: The criteria for a drug resistance mutation was having two consecutive visits of HBV DNA ≥ 69 IU/mL.
Time Frame: Baseline up to Week 48
Population: There were no participants analyzed for the outcome measure since none of the participants met the criteria.
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (maximum duration: 24 Weeks) plus 30 days; All Cause Mortality: Randomization up to 28 months
Description: Adverse Events: The Safety Analysis Set included all randomized participants who took at least 1 dose of the study drug.
  All Cause Mortality: All Randomized Analysis Set includes all participants who were randomized in the study.
Arm/Group | Selgantolimod 3 mg: HBeAg-positive CHB Participants | Selgantolimod 3 mg: HBeAg-negative CHB Participants | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants | Placebo: HBeAg-positive CHB Participants | Placebo: HBeAg-negative CHB Participants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/10 | 0/10 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/10 | 1/10 | 2/10 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10 | 8/10 | 10/10 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selgantolimod 3 mg: HBeAg-positive CHB Participants (N=9) | Selgantolimod 3 mg: HBeAg-negative CHB Participants (N=10) | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants (N=10) | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants (N=10) | Placebo: HBeAg-positive CHB Participants (N=5) | Placebo: HBeAg-negative CHB Participants (N=4)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selgantolimod 3 mg: HBeAg-positive CHB Participants (N=9) | Selgantolimod 3 mg: HBeAg-negative CHB Participants (N=10) | Selgantolimod 1.5 mg: HBeAg-positive CHB Participants (N=10) | Selgantolimod 1.5 mg: HBeAg-negative CHB Participants (N=10) | Placebo: HBeAg-positive CHB Participants (N=5) | Placebo: HBeAg-negative CHB Participants (N=4)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Borderline glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Optic disc disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pinguecula (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 3 | 4 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 2 | 2 | 0 | 1 | 1 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 5 | 1 | 2 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 4 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Citrate toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Urine output increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 2 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 3 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03491553/Prot_000.pdf
  • Statistical Analysis Plan: Week 24 Analysis and Final Analysis (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03491553/SAP_001.pdf
  • Statistical Analysis Plan: TFFU (Treatment-Free Follow-Up) Analysis (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03491553/SAP_002.pdf